CLINICAL TRIAL: NCT05573828
Title: Usefulness of ICG Angiography-Guided Thyroidectomy for Preserving Parathyroid Function. GuiArte Multicentric Randomized Study.
Brief Title: Usefulness of ICG Angiography-Guided Thyroidectomy for Preserving Parathyroid Function
Acronym: GuiArte
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Universitari de Bellvitge (Other)
Responsible Party: Principal Investigator, Pablo Moreno Llorente, Head of Endocrine Surgery, Hospital Universitari de Bellvitge
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: PR161/21
Record Dates: First submitted 2022-10-06; First posted 2022-10-10 (Actual); Last update posted 2025-03-19 (Actual); Status verified 2025-03

CONDITIONS: Iatrogenic Hypocalcemia
Keywords: hypocalcemia; ICG angiography; Guided thyroidectomy
MeSH Terms: conditions — Hypocalcemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Angiography group (Experimental): Patients undergoing initially ICG angiography guided thyroidectomy to identify the vessels feeding the parathyroid glands and then, post-thyroidectomy ICG angiography to predict immediate parathyroid function.
  Interventions: Procedure: ICG angiography to show vascular map of parathyroid glands
- Control group (No Intervention): Patients who underwent post-thyroidectomy ICG angiography to predict immediate parathyroid gland function by scoring the degree of fluorescence of the parathyroid glands

INTERVENTIONS:
Procedure: ICG angiography to show vascular map of parathyroid glands — Using ICG angiography guided thyroidectomy to identify the vessels feeding the parathyroid glands and then perform the thyroidectomy. After it, ICG angiography is done to predict immediate parathyroid functio
  Arms: Angiography group

SUMMARY:
Transient and/or permanent hypoparathyroidism is the most frequent complication after total thyroidectomy. The identification of the parathyroid glands and a correct dissection during thyroidectomy have been postulated as key factors for their preservation and, consequently, to prevent hypoparathyroidism. The use of indocyanine green (ICG) fluorescence has reliably predicted parathyroid glands functionality in the immediate postoperative period. Recently, it is proposed that showing the vascular map of the parathyroid glands before performing the thyroidectomy by means of ICG angiography prevent the development of postoperative hypoparathyroidism.

The goal of this multicentric study is to demonstrate that the preservation of the function of parathyroid glands is greater with use of arteriography than without.

Patients will be divided in two groups. In the study group, the vascular map with ICG of parathyroid glands will be showed before performing the lobectomy. Once the lobectomy is done, the function of the glands will be assessed. Whereas in the control group, arteriography with ICG will only be carried out in order to check their function at the end of the lobectomy.

Researchers will compare the study group and the control group to see which one present the lowest taxes of postoperative hypoparathyroidism.

DETAILED DESCRIPTION:
To assess the appearance of postoperative hypoparathyroidism, a systematic determination of PTH and corrected calcium values will be carried out the morning after the intervention.

It will be considered that there is hypoparathyroidism when the patient presents symptoms of hypocalcaemia, when he has required the administration of calcium and/or vitamin D prior to this determination or when he presents corrected calcium values < 1.8 mmol/L.

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥ 18 years of age with a surgical indication for total thyroidectomy with or without central cervical lymph node dissection due to thyroid pathology.
* The patient or their guardian, where applicable, has the capacity to understand the study and agrees to participate in it, signing the corresponding informed consent document.

Exclusion Criteria:

* Previous surgical intervention on the thyroid or parathyroid gland.
* Associated hyperparathyroidism that requires associating a parathyroidectomy in the same surgical act.
* Patients with contraindications for the administration of ICG.
* Current drug use or alcohol abuse that could interfere with compliance with the study requirements.
* Participation in any other drug trials in the month prior to randomization.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 394 (Estimated)
Dates: Start 2022-10-11 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Rate of participants with postoperative permanent hypoparathyroidism | 1 year
  Comparison of postoperative permanent hypoparathyroidism between the two groups. It is considered permanent hypoparathyroidism in the presence of symptoms of hypocalcemia or less than 1.8mmol/L of calcium in asymptomatic patients during more than 12 months.

SECONDARY OUTCOMES:
Rate of participants with severe permanent hypocalcemia | 1 year
  Comparison of the occurrence of severe permanent hypocalcemia after total thyroidectomy between the two groups. Severe hypocalcemia is considered when vitamin D is added to the treatment with calcium. Permanent hypocalcemia is defined when it lasts more than 12 months.
Number of parathyroid glands identified and preserved | 1 year
  Comparison of the number of parathyroid glands identified, left in situ and with an ICG score of 2 after total thyroidectomy between the two groups.

CONTACTS AND LOCATIONS:
Overall Officials: Pablo Moreno, Principal Investigator — Hospital Universitari de Bellvitge
Locations (2):
- Spain (2):
  - Hospital UIniversitari de Bellvitge, L'Hospitalet de Llobregat, Barcelona
  - Pablo Moreno Llorente, L'Hospitalet de Llobregat, Barcelona

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Edafe O, Antakia R, Laskar N, Uttley L, Balasubramanian SP. Systematic review and meta-analysis of predictors of post-thyroidectomy hypocalcaemia. Br J Surg. 2014 Mar;101(4):307-20. doi: 10.1002/bjs.9384. Epub 2014 Jan 9. PMID 24402815
- [Background] Vidal Fortuny J, Sadowski SM, Belfontali V, Karenovics W, Guigard S, Triponez F. Indocyanine Green Angiography in Subtotal Parathyroidectomy: Technique for the Function of the Parathyroid Remnant. J Am Coll Surg. 2016 Nov;223(5):e43-e49. doi: 10.1016/j.jamcollsurg.2016.08.540. Epub 2016 Aug 24. No abstract available. PMID 27568330
- [Background] Falco J, Dip F, Quadri P, de la Fuente M, Prunello M, Rosenthal RJ. Increased identification of parathyroid glands using near infrared light during thyroid and parathyroid surgery. Surg Endosc. 2017 Sep;31(9):3737-3742. doi: 10.1007/s00464-017-5424-1. Epub 2017 Mar 31. PMID 28364157
- [Background] Benmiloud F, Penaranda G, Chiche L, Rebaudet S. Intraoperative Mapping Angiograms of the Parathyroid Glands Using Indocyanine Green During Thyroid Surgery: Results of the Fluogreen Study. World J Surg. 2022 Feb;46(2):416-424. doi: 10.1007/s00268-021-06353-4. Epub 2021 Nov 6. PMID 34743241
- [Background] Llorente PM, Francos Martinez JM, Barrasa AG. Intraoperative Parathyroid Hormone Measurement vs Indocyanine Green Angiography of Parathyroid Glands in Prediction of Early Postthyroidectomy Hypocalcemia. JAMA Surg. 2020 Jan 1;155(1):84-85. doi: 10.1001/jamasurg.2019.3652. PMID 31617879
- [Result] Moreno-Llorente P, Garcia-Barrasa A, Pascua-Sole M, Videla S, Otero A, Munoz-de Nova JL. Usefulness of ICG Angiography-Guided Thyroidectomy for Preserving Parathyroid Function. World J Surg. 2023 Feb;47(2):421-428. doi: 10.1007/s00268-022-06683-x. Epub 2022 Aug 9. PMID 35945357
- [Derived] Moreno-Llorente P, Garcia-Gonzalez G, Pascua-Sole M, Garcia-Barrasa A, Videla S, Munoz-de-Nova JL; GuiArte Study Group. Indocyanine green angiography-guided thyroidectomy versus conventional thyroidectomy for preserving parathyroid function: study protocol for a randomized single-blind controlled trial. Front Endocrinol (Lausanne). 2023 May 8;14:1193900. doi: 10.3389/fendo.2023.1193900. eCollection 2023. PMID 37223015